CLINICAL TRIAL: NCT05391724
Title: An Open-Label Study to Determine the Safety and Pharmacokinetics of CMX001 in Subjects With Impaired Hepatic Function and Healthy Subjects With Normal Hepatic Function
Brief Title: Safety and Pharmacokinetics of CMX001 in Impaired Hepatic Function and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMX001-106
Record Dates: First submitted 2011-06-30; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hepatic Impairment
Keywords: hepatic impairment
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMX001 (Experimental): single dose of CMX001 administered at 2 mg/kg of ideal body weight rounded to the closest 20 mg
  Interventions: Drug: CMX001

INTERVENTIONS:
Drug: CMX001 — single dose of CMX001 administered at 2 mg/kg of ideal body weight rounded to the closest 20 mg
  Other Names: Brincidofovir; BCV

SUMMARY:
This is an open-label, non-randomized, multi-center, sequential group, safety, tolerance, and Pharmacokinetic study of a single dose of CMX001 administered at 2 mg/kg of ideal body weight rounded to the closest 20 mg in fasted healthy control subjects compared with that in fasted subjects with moderate and severe hepatic impairment.

DETAILED DESCRIPTION:
A maximum of 24 subjects will be studied at multiple sites in the Unites States. Eight subjects with normal hepatic function and 8 subjects with moderate hepatic impairment will be enrolled on Cohort 1 and an additional 8 subjects with severe hepatic impairment may be enrolled in Cohort 2. The severity of hepatic impairment will be assessed according to the Child-Pugh-Turcotte (CPT) score1 (see Table 4-2). Because CMX001 is highly protein-bound, to avoid confounding the PK assessment of hepatic impairment versus hypoalbuminemia, only patients with serum albumin levels >3 g/dL will be enrolled in this study.

Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to Check-in.

Subjects who have met inclusion and exclusion criteria will check in to the clinic on Day -1 and receive a single oral dose of CMX001 (2 mg/kg of ideal body weight rounded to the closest 20 mg) on Day 1. The study design schematic is presented in Table 4-3. Subjects will be discharged from the clinic on Day 2 (if stable in the opinion of the Investigator), return for outpatient visits on Days 3 through 6 for safety assessments and PK sampling, and return for an End of Study Visit on Day 14 ± 2 for safety assessments. Subjects may be confined to the clinic during the period of Day -1 to Day 6 at the discretion of the Investigator, after discussion with the Medical Monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF);
2. Male or female subjects, between 18 and 65 years of age, inclusive;
3. Within body mass index (BMI) range 18 to 40 kg/m2, inclusive;
4. Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (does include alcohol); positive drug screens in the hepatically-impaired subjects may be allowed with the confirmation of use of the medication under supervision of a physician)
5. Negative HIV antibody and hepatitis B surface antigen (HBsAg) screens;
6. Female subjects will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year (with follicle-stimulating hormone (FSH) levels ≥40 mIU/mL), surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days, or agree to use from the time of signing the ICF until 30 days after Study Discharge one of the following forms of contraception: a non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; a non-hormonal intravaginal system; diaphragm with spermicide; cervical cap with spermicide; a male sexual partner who agrees to use a male condom with spermicide; or a sterile sexual partner; for all female subjects, the pregnancy test result must be negative at Screening and Check-in;
7. Male subjects will either be sterile or agree to use from Check-in until 45 days following Study Discharge one of the following approved methods of contraception: a male condom with spermicide; a sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; an intravaginal system (e.g., NuvaRing®); a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives.

For healthy subjects with normal hepatic function:

1. Normal hepatic function defined as alanine aminotransferase, aspartate aminotransferase, bilirubin, serum albumin, and gamma glutamyl transferase all within normal limits;
2. The absence of clinically-relevant abnormalities identified by a detailed medical history, full physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests;
3. Negative hepatitis panel (including HBsAg and hepatitis C virus antibody);
4. No medical or surgical conditions that might significantly interfere with gastrointestinal absorption of CMX001.

For subjects with impaired hepatic function:

1. Otherwise healthy subjects as determined by a detailed medical history, complete physical examination, vital signs, 12-lead ECG, and clinical laboratory tests (abnormal findings that are related to the subject's underlying condition are acceptable);
2. Satisfy the criteria for Class B or Class C of the modified Child-Turcotte-Pugh (CPT) classification (mild [CPT score of 5 to 6 points], moderate [CPT score of 7 to 9 points], and severe [CPT score of >9 to <12 points]);
3. A diagnosis of chronic hepatic impairment due to cirrhosis or fibrosis, not secondary to other diseases, which is confirmed and documented by medical history, physical examination, and/or liver biopsy, hepatic ultrasound, computed tomography scan, or magnetic resonance imaging.

Exclusion Criteria:

1. Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic (healthy control subjects only), renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator, Sponsor, and/or Sponsor's representative);
2. Any non-hepatic disease or condition that could affect safety or data interpretation (as determined by the Investigator, Sponsor, and/or Sponsor's representative);
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, including cidofovir (CDV), food, or other substance, unless approved by the Investigator, Sponsor, and/or Sponsor's representative;
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and/or hernia repair will be allowed;
5. History of any condition possibly affecting drug absorption (e.g., gastrectomy, active peptic ulcer) within the last 3 months;
6. serum albumin <3 g/dL;
7. History or presence of an abnormal ECG, which, in the opinion of the Investigator, Sponsor, and/or Sponsor's representative, is clinically significant;
8. History of alcoholism or drug addiction within 1 year prior to Check-in (healthy control subjects only);
9. Use of any tobacco- or nicotine-containing products within 6 months prior to Check-in (healthy control subjects only);
10. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days (or 5 half-lives, whichever is longer) prior to Check-in;
11. Use of oral, implantable, injectable, or transdermal contraceptives within 14 days prior to Check-in (female subjects only);
12. For healthy control subjects, use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator and Sponsor;
13. For healthy control subjects, use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic/ herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator, Sponsor, and/or Sponsor's representative;
14. Use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours prior to Check-in, unless deemed acceptable by the Investigator, Sponsor, and/or Sponsor's representative;
15. Poor peripheral venous access;
16. Donation of blood during the period of 30 days prior to Screening or donation of plasma during the period of 2 weeks prior to Screening;
17. Receipt of blood products within 2 months prior to Check-in;
18. Any acute or chronic non-hepatic condition that, in the opinion of the Investigator, Sponsor, and/or Sponsor's representative, would limit the subject's ability to complete and/or participate in this clinical study;
19. History of liver transplant;
20. History of febrile illness within 5 days prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 6 months
  An objective of this study was to determine the safety following administration of a single dose of CMX001 in subjects with moderate and severe hepatic impairment compared to match subjects with normal hepatic function.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of moderate and severe hepatic impairment after a single dose of CMX001 | 6 months
  An objective of this study was to evaluate the effects of moderate and severe hepatic impairment on the pharmacokinetic (PK) parameters for CMX001 after a single dose, including Cmax.
Time to maximum concentration (Tmax) of moderate and severe hepatic impairment after a single dose of CMX001 | 6 months
  An objective of this study was to evaluate the effects of moderate and severe hepatic impairment on the pharmacokinetic (PK) parameters for CMX001 after a single dose, including Tmax.
Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) of moderate and severe hepatic impairment after a single dose of CMX001 | 6 months
  An objective of this study was to evaluate the effects of moderate and severe hepatic impairment on the pharmacokinetic (PK) parameters for CMX001 after a single dose, including AUCinf.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Elite Research, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota